CLINICAL TRIAL: NCT03375593
Title: Narcotic Versus Non-narcotic Medication for Pain Management After Wrist/Hand Fractures: a Randomized Controlled Trial
Brief Title: Narcotic Versus Non-narcotic Medication for Pain Management After Wrist/Hand Fractures
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REB 1090503
Record Dates: First submitted 2017-09-05; First posted 2017-12-18 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Distal Radius Fracture; Pain Management; Metacarpal Fracture
Keywords: pain management; RCT
MeSH Terms: conditions — Wrist Fractures; Agnosia | interventions — Hydrocodone; Acetaminophen; Oxycodone; Ibuprofen

STUDY DESIGN:
Intervention Model Description: participants will be randomized to receive either the narcotic hydrocodone with acetaminophen or a combination of acetaminophen plus ibuprofen for post-fracture pain
Who Masked: Participant, Investigator
Masking Description: study medication will be masked to participant and investigator. Medication will be dispensed by pharmacy in identical blister packs
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Narcotic (Experimental): Hydrocodone 5mg/Acetaminophen 500 mg Tab
  Interventions: Drug: Acetaminophen 500Mg Tab; Drug: Ibuprofen 600 mg tab
- Non Narcotic (Experimental): Ibuprofen 600mg Tab + acetaminophen 500 mg Tab
  Interventions: Drug: Hydrocodone 5Mg/Acetaminophen 500Mg Tab

INTERVENTIONS:
Drug: Hydrocodone 5Mg/Acetaminophen 500Mg Tab — tablet
  Other Names: oxycodone
  Arms: Non Narcotic
Drug: Acetaminophen 500Mg Tab — tablet
  Other Names: tylenol
  Arms: Narcotic
Drug: Ibuprofen 600 mg tab — tablet
  Other Names: advil
  Arms: Narcotic

SUMMARY:
The purpose of this study is to evaluate two drug options for pain control in patients following wrist injury. Participants will be randomized to one of the 2 pain relief treatments to determine what treatment provides the most effective pain relief

DETAILED DESCRIPTION:
The purposes of this noninferiority randomized clinical trial are to determine whether: 1. the most commonly used non-narcotic analgesic (ibuprofen 600 mg + acetaminophen 500 mg) provides pain relief that is not unacceptably worse than the most commonly prescribed narcotic (hydrocodone 5 mg + acetaminophen 500 mg) in patients with a hand or wrist fracture. 2. the following covariates affect pain outcomes: sex/gender, age, gender-related pain expectations, paid/unpaid work roles, comorbid health status, baseline pain intensity, and employment status.

ELIGIBILITY:
Inclusion Criteria:

* All patients 18 and older undergoing non-operative management of a hand or wrist fracture will be considered eligible.
* Able to read and speak English

Exclusion Criteria:

* pain exceeding 7/10 on numeric rating scale or 35/50 on PRWE pain scale at enrollment
* nerve injury
* surgeon decision that surgery is required
* history of chronic opioid use
* documented or suspected substance abuse
* individuals currently on daily use of ibuprofen, acetaminophen or other pain-altering medication including medications like Neurontin (gabapentin) and Ultram (tramadol)
* individuals with documented or suspected chronic pain syndrome, reported allergy or adverse reaction to hydrocodone, acetaminophen, or ibuprofen
* history or symptoms of serious medical problem in the last year (i.e., arrhythmia, impaired cardiovascular function, gastrointestinal bleeding, liver disease, renal disease)
* patients with active peptic ulcer disease (history of severe heartburn)
* symptoms of infection
* pregnant or lactating women
* diagnosis of cognitive impairment
* unable to provide informed consent
* unable or unwilling to fill out the forms
* prior fracture in same hand
* on Coumadin or Plavix
* other medical or psychological health conditions that preclude them from receiving either intervention
* or unable to return for follow-up visits

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Pain | 0-2 weeks
  PRWE (patient rated wrist evaluation)
  1. Pain subscale: contains 5 items each of which is further rated from 1-10. The maximum score in this section is 50 and minimum 0
  2. Function subscale: contains total 10 items which are further divided into 2 sections i.e specific activities (having 6 items) and usual activities (having 4 items). The maximum score in this section is 50 and minimum 0

SECONDARY OUTCOMES:
Drug use | 2 weeks
  Total medication used will be recorded by a pain diary (for the first 2 weeks)
Pain diary | 2 weeks
  participants will be provided a pain diary (for the first 2 weeks) that includes the numeric pain rating scale (NRS), where they can record when they take their medication and the NRS at each self-administration. will use a 0-10 scale where 0 means no pain and 10 is the worst imaginable pain
Grip strength | 12 weeks
  Grip strength in kg will be measured with calibrated instrument and standardized test positioning.
Grip strength | 24 weeks
  Grip strength in kg will be measured with calibrated instrument and standardized test positioning.
Pinch strength | 12 weeks
  pinch strength in kg will be measured with calibrated instrument and standardized test positioning.
Pinch strength | 24 weeks
  pinch strength in kg will be measured with calibrated instrument and standardized test positioning.
Dexterity | 12 and 24 weeks
  dexterity will be tested with a standardized test. dexterity is a timed, in seconds, test. the participant is asked to move small objects from one spot to another.
Range of Motion | 12 and 24 weeks
  active range of motion will be measured in degrees with standardized test positioning.
pain management | 3 weeks
  Patient satisfaction with pain management will be measured using a single item satisfaction NRS. using a 0-10 scale where 0 is very unsatisfied and 10 is very satisfied
Work Impact | 12 and 24 weeks
  Time to return to work will be collected and the Work Limitations Questionnaire will be administered at return to work, 12 and 24 weeks to determine the work impacts of interventions. Scale scores range from 0 (limited none of the time) to 100 (limited all of the time)
Future preference | 24 weeks
  Preference for future pain management. Patients will be asked if they were to have another fracture, would they prefer to have the same or a different pain medication. They will also be asked what medication they thought they were taking so we can assess how this impacts on their preference, and to discern whether patients were aware of their allocation
Adverse events | 24 weeks
  Adverse events or complications will be recorded using a standardized complications checklist and a standardized adverse event reporting form completed by their surgeon at each time point

CONTACTS AND LOCATIONS:
Overall Officials: Joy C MacDermid, PhD, Principal Investigator — St. Joseph's Health Care London
Locations (1):
- St. Joseph Health Care, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
only de-identified data will be available upon request